CLINICAL TRIAL: NCT01995786
Title: Clinical Outcomes and Costs Analyses in Use of Goal Directed Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, chief, Regina Elena Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 19.11
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Postoperative Complications
Keywords: Fluid Therapy; Cost-Benefit Analysis; Hemodynamics; Cost Control
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Intravenous Fluid therapy (No Intervention): Basal infusion of crystalloid (normal saline,Ringer's lactate,Ringer's solution)variable from 4 to 12 ml/kg/hour
- GDT (Experimental): Basal infusion of crystalloids (normal saline,Ringer's lactate,Ringer's solution) at 2,5 ml/kg/h and boluses of crystalloids for values of stroke volume (SV) < SV TRIGGER. Every additional infusion of colloids, blood derivates, drugs must be recorded
  Interventions: Device: Goal Directed Fluid Therapy FloTrac/Vigileo

INTERVENTIONS:
Device: Goal Directed Fluid Therapy FloTrac/Vigileo
  Arms: GDT

SUMMARY:
The aim of the study is to evaluate clinical and economic impact of Goal Directed Fluid Therapy according to NICE haemodynamic protocol. Haemodynamic parameters were assessed using automated pulse contour analysis (Flotrac/Vigileo®). A specific dedicated software has been developed to perform clinical and expenditures data collection, both retrospective and prospective data are archived.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for major abdominal surgery

Exclusion Criteria:

•Patients under the age of 18, patients with hemodynamically significant aortic regurgitation and heart rhythm disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
rate of reduction of postoperative spending | 30 day postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ester Forastiere, Principal Investigator — Regina Elena CI
Locations (1):
- Regina Elena CI, Rome, Italy, Italy